CLINICAL TRIAL: NCT05703815
Title: EpCAM and p53 Expressions in Infiltrating Duct Carcinoma of the Breast and Their Association With the Clinicopathological Prognostic Paremeters
Brief Title: EpCAM and p53 Expressions in Infiltrating Duct Carcinoma of the Breast
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rasha Mokhtar Abdelkareem, lecturer, Sohag University
Other Study IDs: Soh-Med-23-01-34
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Invasive Breast Cancer
Keywords: EpCAM, P53 , IDC
MeSH Terms: conditions — Colorectal Cancer, Hereditary Nonpolyposis, Type 8

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer represents the most frequently diagnosed cancer in women. It represents the 5th leading cause of cancer mortality all over the world.

In Egypt, breast cancer represents the 2nd most diagnosed cancer among all population. But among Egyptian females it represents the 1st diagnosed cancer representing 32.4%.

The main cause of death in breast cancer patients is tumor metastasis. Although only 5-10% of recently diagnosed breast cancer cases show metastasis to distant sites, but still there is a high risk for metastasis in patients with localized primary tumor following successful surgical management.

Epithelial cell adhesion molecule (EpCAM) is a cell adhesion molecule. It modifies cadherin mediated cell adhesion and it induces epithelial cell migration and proliferation. Some authors elucidate that EpCAM is involved in metastasis.

P53 is a known tumor suppressor gene involved in the control of cell cycle, DNA repair and apoptosis. It's one of the most mutated genes in cancer including breast cancer. Mutant p53 has a big role in tumor progression.

ELIGIBILITY:
Inclusion Criteria:

- Both incisional and excisional biopsy specimens. 2. All the studied cases include sufficient materials for the immunohistochemical study.

3. Complete clinical data.

Exclusion Criteria:

1. Patients with recurrence of the primary tumor.
2. Patients with a history of preoperative chemotherapy and/or radiotherapy.
3. Insufficient or tiny tissue biopsies

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: formalin-fixed and paraffin embedded tissue blocks from 40 patients with breast cancer
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of breast cancer | two day after staining sections with Immnnohistochemical markers
  Immunohistochemical expression of EpCAM and P53 in IDC of the breast

CONTACTS AND LOCATIONS:
Overall Officials: Rasha M Abdelkareem, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: Undecided